CLINICAL TRIAL: NCT00576511
Title: A Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of R093877 in Patients With Severe Chronic Constipation
Brief Title: Effect of Prucalopride in Patients With Severe Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-BEL-6
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2007-12

CONDITIONS: Chronic Constipation
Keywords: Constipation; Prucalopride; Colonic Transit Time
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Prucalopride
  Interventions: Drug: prucalopride
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prucalopride — 4 mg o.d.
  Other Names: Resolor
  Arms: 1
Drug: placebo — Placebo o.d.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether prucalopride is safe and effective in patients with severe chronic constipation.

DETAILED DESCRIPTION:
This is a phase II trial with a parallel-group design, consisting of a run-in phase (phase I), followed by a placebo controlled double-blind phase (phase 2). Patients will receive either R093877 4 mg or placebo o.d. for a period of 4 weeks.

Phase 1 is a run-in period of 4 weeks duration, during which the bowel habit is documented and the existence of constipation determined. If the definition of constipation was not met during the 4 weeks of the run-in period, double-blind treatment will not be started.

Phase 2 is a double-blind, randomized, placebo-controlled phase, in which patients will be treated for 4 weeks with either 4 mg of R093877 or placebo given o.d. (two capsules of 2 mg are taken before breakfast).

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were aged 18-75 years with a history of constipation, defined as the occurrence 2 of the following criteria during the previous 6 months or more:

  * 2 spontaneous (i.e. not induced by a laxative within 24 hours) bowel movements per week;
  * 25% of stools were lumpy and/or hard;
  * sensation of incomplete evacuation following 25% of stool;
  * straining at defaecation for 25% of the time.

All the patients screened for the study were dependent on osmotic laxatives (macrogol, milk of magnesia, lactulose), paraffin oil, glycerol or stimulant laxatives (antranoids, diphenylmethanes) given orally or rectally. The osmotic laxatives were taken on a daily base while the stimulant laxatives were restricted to 2, eventually 3 intakes per week. And although these laxatives, all or not combined promoted defaecation in the majority of patients, these regimens did not provide relief of constipation symptoms in none of the patients. Furthermore, many patients reported that the effect of the laxatives declined over time, that the intake of even stimulant laxatives was not consistently followed by rectal evacuation or that the intake of even stimulant laxatives was not consistently followed by rectal evacuation of that the dose and frequency of intake of laxatives had to be limited because of intolerable side effects including vomiting and abdominal cramps.

Eligible patients were also required to have constipation causing disability, with the patient's occupational, social and recreational activities governed by constipation and efforts to attain relief, and to have poor results with laxative treatment and diet counseling as determined by physician interview.

Patients also had to have a normal electromyographic inhibition pattern of the external anal sphincter during straining (assessed at the start of the treatment phase) and an absence of organic abnormalities of the colon (as assessed by barium enema or total colonoscopy).

Exclusion Criteria:

* Drug-induced constipation
* Secondary causes of constipation
* Known or suspected organic large bowel disorders
* Congenital or acquired megacolon/megarectum
* History of previous abdominal surgery
* Evidence of a non-relaxing pelvic floor as the main cause of constipation
* Active proctological conditions
* Impaired renal function or clinically significant abnormalities of blood chemistry, hematology, urinalysis or ECG.
* Patients who were pregnant, breast feeding, not using acceptable methods of birth control or who had known illnesses or conditions that might interfere with adequate assessment of the study drug were also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1994-12; Primary Completion 1996-02 (Actual); Study Completion 1996-02 (Actual)

PRIMARY OUTCOMES:
Constipation severity (VAS) | 4 weeks

SECONDARY OUTCOMES:
Stool frequency (stool/week) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georges Coremans, MD, Principal Investigator — Department of Gastroenterology, University Hospital Gasthuisberg, Catholic University Leuven, Leuven

REFERENCES:
- [Result] Coremans G, Kerstens R, De Pauw M, Stevens M. Prucalopride is effective in patients with severe chronic constipation in whom laxatives fail to provide adequate relief. Results of a double-blind, placebo-controlled clinical trial. Digestion. 2003;67(1-2):82-9. doi: 10.1159/000070202. PMID 12743445